CLINICAL TRIAL: NCT02124473
Title: Phase II Randomized, Double-Blind, Placebo-Controlled Trial of Homeopathy in Resistant Arterial Hypertension
Brief Title: Addition of Homeopathy in Patients With Resistant Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mac/NMP 1120
Record Dates: First submitted 2014-04-20; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Resistant hypertension; Homeopathy; Blood pressure; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy | interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homeopathy (Experimental): A range of homeopathic potencies were used as per the individualized requirement, decided by the treating physicians.Each dose, administered orally, (in centesimal potencies).
  Interventions: Other: Homeopathy
- Placebo (Placebo Comparator): Placebo, identical in appearance, consisted of 83.1% ethanol in 10 ml distilled water and was served in identical amber-coloured glass vials
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Homeopathy
  Arms: Homeopathy
Other: Placebo
  Arms: Placebo

SUMMARY:
Resistant hypertension (RHTN) is a common clinical problem faced by both primary care clinicians and specialists worldwide. Patients with RHTN have higher rates of cardiovascular events and mortality compared with patients with more easily controlled hypertension. In addition, RHTN is often complicated by metabolic abnormalities.

Homeopathy, although widely used in hypertension, but no study has been taken to evaluate the impact on resistant hypertension. The aim of this trial was to evaluate individualized homeopathy on BP in patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with resistant arterial hypertension.
* Office systolic BP >140 mm Hg or diastolic BP >90 mm Hg despite being treated with at least 3 antihypertensive drugs, including a diuretic.
* Patients with diabetes or chronic kidney disease (defined as serum creatinine >133 μmol/L or proteinuria >300 mg/day) if the office BP was >130/80 mm Hg.

Exclusion Criteria:

* Severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg) who needed an immediate adjustment of treatment,
* Renal insufficiency with serum creatinine >180 μmol/L or glomerular filtration rate <40 mL/min calculated by the Modification of Diet in Renal Disease formula,15 hyperkalemia >5.4 mmol/L, hyponatremia <130 mmol/L, and porphyria;
* Pregnant or lactating women or women of fertile age not using effective contraception;
* Patients with known prior hypersensitivity to the drug Verospiron (spironolactone; Richter Gedeon Ltd) or who are currently using any aldosterone antagonist.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Daytime systolic and diastolic pressure | Change from Baseline in Systolic and Diastolic Blood Pressure at 3 months

SECONDARY OUTCOMES:
24-hour systolic and diastolic BP | Change from Baseline in 24-hour blood pressure at 3 months

OTHER OUTCOMES:
Serum levels of sodium | Change from Baseline in Serum level of sodium at 3 months
Serum levels of potassium | Change from Baseline in serum levels of potassium at 3months
Serum levels of creatinine | Change from Baseline in Serum levels of creatinine at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vipin Sharma, BHMS, Principal Investigator — NMP Medical Research Institute, India; Neha Sharma, Study Director — Macmillan Research Group UK
Locations (2):
- India (2):
  - NMP Medical Research Institute, Jaipur, Rajasthan
  - NMP Medical Research Institute, Jhunjhunūn, Rajasthan